CLINICAL TRIAL: NCT06328608
Title: Multi-centre, Open-label Trial to Assess the saFety, Pharmacodynamics, Efficacy and Pharmacokinetics of pegunigaLsidase Alfa in Patients From 2 Years to Less Than 18 Years of Age With Confirmed FabrY Disease
Brief Title: A Study to Learn About the Safety and Effects of the Study Drug PRX-102 in Children and Adolescents With Fabry Disease
Acronym: FLY
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLI-06657AA1-01; 2022-503128-29 (Registry Identifier: Clinical Trial Information System (CTIS) - EU)
Record Dates: First submitted 2023-08-10; First posted 2024-03-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm - Pegunigalsidase alfa (PRX-102) (Experimental): For Cohort C, PXR-102 administered every two weeks at 1.0 mg/kg is believed to be the minimum effective dose.
  For Cohorts A and B, the starting dose will be 1.0 mg/kg every two weeks but it may be adjusted on the outcomes of Stage I, with the support of the Data Safety Monitoring Board.
  Interventions: Drug: PRX-102 1 mg/kg every two weeks

INTERVENTIONS:
Drug: PRX-102 1 mg/kg every two weeks — Drug: PRX-102 1 mg/kg every two weeks
  Other Names: pegunigalsidase alfa; Recombinant human alpha galactosidase-A

SUMMARY:
A Study to Learn About the Safety and Effects of the Study Drug PRX-102 in Children and Adolescents with Fabry Disease.

DETAILED DESCRIPTION:
This study aims to learn how safe pegunigalsidase alfa (PRX-102 for short) is and how it works at treating Fabry disease in children and adolescents.

PRX-102 is an enzyme replacement therapy (ERT), meaning it acts like a natural enzyme. PRX-102 is given through a needle placed in a vein (intravenous infusion) every two weeks.

The main questions this study aims to answer are:

* Which is the safest and most effective dose to be given to children and adolescents.
* Which effects PRX-102 has on signs and symptoms of Fabry disease (e.g. renal and cardiac function, pain, gastrointestinal symptoms)

  20 to 22 boys and girls with Fabry disease between the ages of 2 and 17 will be part of this study. There will be three age cohorts, with children aged 2 to 7 years included (enrolled) in Cohort A, children aged 8 to 12 years in Cohort B, and adolescents aged 13 to less than 18 years in Cohort C.

The study is divided into three parts, or "stages":

* A dose-finding stage (Stage I). In this stage, researchers will determine the dose for children.
* A confirmatory stage (Stage II). In this part, researchers will learn about the safety and efficacy of PRX-102.
* and an optional extension stage (Stage III) will continue until the study drug becomes commercially available or the Sponsor chooses to end this study.

PRX-102 will be given at the study visits, which will occur at least every two weeks. Tests for verifying the study drug's safety and efficacy and determining the dose will also be conducted at different time points throughout the study (not all tests will be done at all visits). These tests may include a review of any health problems and medications the participants have had or taken since the last visit; a physical examination; ECG; ultrasound of the heart; questionnaires that evaluate the nature and severity of Fabry disease symptoms, quality of life and pain; a collection of blood and urine samples for standard safety tests, to analyse the severity of Fabry disease and to see how the drug is behaving and how long it remains active in the body (this involves taking multiple blood samples over several days with the first sample taken just before the start of the PRX-102 infusion and the last one taken just before the start of the next PRX-102 at the next visit).

ELIGIBILITY:
Inclusion Criteria:

* Participants with the provision of informed consent from their legal guardians
* Boys and girls aged 2 to 7 years (Cohort A), 8 to 12 years (Cohort B), or 13 to <18 years (Cohort C).
* Confirmed diagnosis of Fabry disease
* Presence of at least one of the following characteristic features of Fabry disease: neuropathic pain, cornea verticillata, and/or clustered angiokeratoma.
* History of Fabry pain: Fabry crises OR chronic pain.
* Clinical condition that, in the investigator's opinion, requires ERT treatment.

Exclusion Criteria:

All Subjects:

* Estimated glomerular filtration rate (eGFR) at screening < 80 mL/min/1.73 m2.
* History of type I hypersensitivity reactions (anaphylactic or anaphylactoid life-threatening reaction) to other ERT treatment for Fabry disease or any component of the study drug.
* Initiation of treatment with an angiotensin-converting enzyme inhibitor (ACEi) or angiotensin II receptor blocker (ARB) or a dose change in ongoing treatment in the four weeks before screening.
* Urine protein to creatinine ratio (UPCR) > 0.5 g/g (0.5 mg/mg or 500 mg/g) if not treated with an ACE inhibitor or ARB.
* Currently taking another investigational drug for any condition.
* History of acute kidney injury in the 12 months before screening, including specific kidney diseases (e.g., acute interstitial nephritis, acute glomerular and vasculitic renal diseases); non-specific conditions (e.g., ischaemia, toxic injury); or extrarenal pathology (e.g., prerenal azotaemia, acute postrenal obstructive nephropathy).
* History of renal dialysis or kidney transplantation.
* History of or current malignancy requiring treatment.
* Severe cardiomyopathy or significant unstable cardiac disease within six months before screening.
* A positive test for Severe Acute Respiratory Syndrome-Coronavirus 2 (SARS-CoV-2) within three months before screening.
* Presence of any medical, emotional, behavioural, or psychological condition that, in the Investigator's judgement, could interfere with the subject's compliance with the requirements of the study.

Additional Exclusion Criteria for Subjects Enrolled in Stage I:

* Female
* Non-classic form of Fabry disease
* Receipt of treatment for Fabry disease within six months before screening
* Positive for anti-PRX-102 antibodies at screening

Additional Exclusion Criteria for Subjects in Stage II (i.e., non-treatment naïve males or females):

* Unwilling to discontinue current ERT treatment for Fabry disease before baseline.
* Females: Pregnant or lactating, or of childbearing potential with a fertile male partner and unwilling to use a highly reliable method of contraception from the informed consent signature until 30 days after the last infusion.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events (TEAEs) | 12 Months
Incidence of Infusion Related Reactions (IRRs) | 12 Months
Incidence of Injection site reactions (ISRs) | 12 Months
Change in Tanner stage | Baseline and 12 Months
  Tanner Staging of Sexual Development will be used to assess sexual development (i.e. breast development (B1 to B5) and pubic hair development (Ph-1 to Ph-5) in females and pubic hair and genetical development (G1-G5) in males.
Change from baseline of 12-lead ECG quantitative parameters: Mean Heart Rate | Baseline and 12 Months
Change from baseline of 12-lead ECG quantitative parameters: PR Interval | Baseline and 12 Months
Change from baseline of 12-lead ECG quantitative parameters: QRS Duration | Baseline and 12 Months
Change from baseline of 12-lead ECG quantitative parameters: QT Interval | Baseline and 12 Months
Change from baseline of 12-lead ECG quantitative parameters: QTc Interval | Baseline and 12 Months
Change from baseline of 12-lead ECG quantitative parameters: ST Segment | Baseline and 12 Months
Incidence of treatment-emergent Anti-Drug Antibodies (ADAs) | Baseline and 12 Months
Incidence of premedication use at each visit and change of infusion premedications from baseline | Baseline and 12 Months
Pharmacokinetics: Time to maximum plasma concentration (tmax) | Stage I - Baseline, week 2, week 4, week 12, week 26 and week 52; Stage II -Baseline, week 12, week 26 and week 52]
Pharmacokinetic : Area under the plasma concentration-time curve from time 0 to time t (AUC0 t) | Stage I - Baseline, week 2, week 4, week 12, week 26 and week 52; Stage II -Baseline, week 12, week 26 and week 52]
Pharmacokinetics: Area under the curve from time 0 to 2 weeks (AUC0-2wk) | Stage I - Baseline, week 2, week 4, week 12, week 26 and week 52; Stage II -Baseline, week 12, week 26 and week 52]
Pharmacokinetics: Area under the curve from time 0 to infinity (AUC0-∞) | Stage I - Baseline, week 2, week 4, week 12, week 26 and week 52; Stage II -Baseline, week 12, week 26 and week 52]
Pharmacokinetics: Terminal half-life (t1/2) | Baseline, week 2, week 4, week 12, week 26 and week 52]
Pharmacokinetics: Area under the curve over a dosing interval (AUCτ) | Baseline, week 2, week 4, week 12, week 26 and week 52; Stage II -Baseline, week 12, week 26 and week 52]
Pharmacokinetics: Observed drug concentration at the end of the dosing interval (Cτ) | Stage I - Baseline, week 2, week 4, week 12, week 26 and week 52; Stage II -Baseline, week 12, week 26 and week 52]
Pharmacokinetics: Clearance (Cl) | Stage I - Baseline, week 2, week 4, week 12, week 26 and week 52; Stage II -Baseline, week 12, week 26 and week 52]
Pharmacokinetics: Volume of distribution (Vz) | Stage I - Baseline, week 2, week 4, week 12, week 26 and week 52; Stage II -Baseline, week 12, week 26 and week 52]
Change in eGFR | Baseline and 12 Months
Change in annualized eGFR slope | Baseline and 12 Months
Change in urine albumin levels | Baseline and 12 Months
Change in urine protein levels | Baseline and 12 Months
Change from baseline in LVMi as assessed by echocardiogram | Baseline and 12 Months
  Echocardiogram parameters include left ventricular mass index (LVMi)
Change from baseline in LVMi as assessed by echocardiogram | Baseline and 12 Months
  Echocardiogram parameters include ejection fraction
Change from baseline in LVMi as assessed by echocardiogram | Baseline and 12 Months
  Echocardiogram parameters include, fractional shortening
Change from baseline in LVMi as assessed by echocardiogram | Baseline and 12 Months
  Echocardiogram parameters include left ventricular mass
Change from baseline in LVMi as assessed by echocardiogram | Baseline and 12 Months
  Echocardiogram parameters include valve abnormalities and thickness.
Incidence of any cardiac arrythmias as assessed by Holter ECG | Baseline and 12 Months
Change in plasma levels of cardiac biomarkers | Baseline and 12 Months
  High-sensitivity cardiac troponin T (hs-cTnT) and N- terminal pro brain natriuretic peptide (NT-Pro BNP) will be assessed.
Change in plasma level of Gb3 concentration (nM) | Baseline and 12 Months
Change in plasma level of lyso-Gb3 (nM) | Baseline and 12 Months
Change in urine level of lyso-Gb3 (nM) | Baseline and 12 Months
Incidence of change from baseline in the number of different pain medications | Baseline and 12 Months
Incidence of Fabry Clinical Events | 12 Months
  FCEs are classified into four categories: renal, cardiac, cerebrovascular and death due to non-cardiac reasons
Change from baseline of Mainz Severity Score Index (MSSI) scores | Baseline and 12 Months
  Domains (general, neurological, cardiovascular, renal dysfunction)
Change from baseline of PedsQL-GI (or GSRS for subjects who reaches 18 yrs of age) scores | Baseline and 12 Months
Change from baseline of FPHPQ scores | Baseline and 12 Months
Change from baseline of PedsQL-PPQ (or BPI-SF for subjects who reaches 18 yrs of age) scores | Baseline and 12 Months
Change from baseline of EQ-5D-Y (or EQ-5D-5L for subjects who reaches 18 yrs of age) scores | Baseline and 12 Months

CONTACTS AND LOCATIONS:
Locations (12):
- United States (6):
  - Phoenix Children's, Phoenix, Arizona
  - Emory Genetics Clinical Trials Center, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Utah, Salt Lake City, Utah
  - Lysosomal and Rare Disorders Research and Treatment Center Inc, Fairfax, Virginia
- UK für Kinder- und Jugendheilkunde der PMU Salzburg, Salzburg, Austria
- France (2):
  - Centre Hospitalier Universitaire (CHU) de Bordeaux - Groupe Hospitalier Pellegrin, Bordeaux
  - Hopital Arnaud de Villeneuve, Montpellier
- Haukeland Universitetssjukehus, Bergen, Norway
- Hospital Clinico Universitario De Santiago De Compostela, Santiago de Compostela, Spain
- Great Ormond Street Hospital for Children NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No